CLINICAL TRIAL: NCT05426317
Title: Study of the Relationship Between the Blood Levels of Soluble PDL1 and β2-microglobulin, and the Clinical Course of a Metastatic Solid Tumor Treated With a First-line Therapeutic of Checkpoint Immune Inhibitor
Brief Title: Exploratory Interventional Study of Prognostic Serum Biomarkers of Cancer Progression
Acronym: Onco-PDL1s/B2M
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2021 DOUGE; 2021-A02495-36 (Other: ANSM)
Record Dates: First submitted 2022-01-14; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-01

CONDITIONS: Melanoma; Non Small Cell Lung Cancer; Renal Cancer
Keywords: imunotherapy; biomarkers; prognostic
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Kidney Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: metastatic solid tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic solid tumor treated with first line therapeutic of Immune Checkpoint Inhibitor (Other): * The determinations of soluble PDL1 and serum B2M will be taken by blood sample at diagnosis and then every 3 months for 1 year, during a consultation or treatment in an outpatient hospital.
  * The measurement of the tumor PDL1 level at diagnosis will be carried out by immunohistochemistry in the anatomopathology department of Clermont Ferrand University Hospital on the tumor sample that allowed the diagnosis, which does not add an additional sample for the patient.
  * Clinical and imaging examinations will be those conventionally carried out in the context of patient monitoring, the data will only be recorded in the patients' medical files.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — This study only involves the patient taking 5 additional blood tests (peripheral venipuncture) compared to his usual care, which will be taken when he comes to the hospital. Each sample only requires a blood volume of 5mL (one tube), or a total blood volume of 25mL for the study (one blood test every 3 months for one year).
  Other Names: Archived tumor sample

SUMMARY:
Exploratory interventional study of prognostic serum biomarkers of cancer progression.

Study of the relationship between the blood levels of soluble PDL1 and β2-microglobulin, and the clinical course of a metastatic solid tumor treated with a first-line therapeutic of checkpoint immune inhibitor.

DETAILED DESCRIPTION:
Primary objective To study the relationship between the blood levels of soluble PDL1 and β2-microglobulin measured at the diagnostic stage, and the clinical course of a metastatic solid tumor (non-small cell lung cancer, kidney cancer, or melanoma) treated with a 1st line therapeutic immune checkpoint inhibitor.

The secondary objectives are:

* To study the relationship between the blood levels of soluble PDL1 and β2-microglobulin measured during treatment, and the clinical course of a metastatic solid tumor treated with a first-line therapeutic immune checkpoint inhibitor.
* To study the correlation between the soluble PDL1 level and the tumor PDL1 level.
* To study the correlation between the blood levels of soluble PDL1 and β2-microglobulin.
* To study the relationship between the blood levels of soluble PDL1 and β2-microglobulin measured during the treatment, and the tolerance of treatment with immune checkpoint inhibitor in 1st line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female, with metastatic cancer of the non-small cell, renal or malignant melanoma type, eligible for treatment with a first-line immune checkpoint inhibitor (immunotherapy alone or in combination with another immunotherapy, chemotherapy or targeted therapy).
* Affiliation to a Social Security organization
* Able to give informed consent to participate in research.

Exclusion Criteria:

* Pregnant women
* Patient under guardianship, curatorship or legal protection
* Patient unable to understand the protocol (language barrier, cognitive difficulties)
* Patient with another active cancer
* Patient with creatinine clearance <60 mL / min
* Patient participating in a therapeutic clinical trial
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
determination of soluble PDL1 | the day of the start of immunotherapy
  ng/mL
determination of soluble B2M | the day of the start of immunotherapy
  mg/L
Imaging tumor response | 3 month after inclusion
  RECIST1.1 criteria
Imaging tumor response | 6 month after inclusion
  RECIST1.1 criteria
Imaging tumor response | 9 month after inclusion
  RECIST1.1 criteria
Imaging tumor response | 12 month after inclusion
  RECIST1.1 criteria

SECONDARY OUTCOMES:
progression-free survival | 6 month after inclusion
  RECIST1.1 criteria
progression-free survival | 12 month after inclusion
  RECIST1.1 criteria
overall survival | 6 month after inclusion
  Alive or Dead
overall survival | 12 month after inclusion
  Alive or Dead
level of tumor PDL1 | CYCLE 1 DAY 1 (each cycle is 21 days)
determination of soluble PDL1 | 3 month after inclusion
  ng/mL
determination of soluble PDL1 | 6 month after inclusion
  ng/mL
determination of soluble PDL1 | 9 month after inclusion
  ng/mL
determination of soluble PDL1 | 12 month after inclusion
  ng/mL
determination of soluble B2M | 3 month after inclusion
  mg/L
determination of soluble B2M | 6 month after inclusion
  mg/L
determination of soluble B2M | 9 month after inclusion
  mg/L
determination of soluble B2M | 12 month after inclusion
  mg/L
adverse events | 3 month after inclusion
  CTCAE
adverse events | 6 month after inclusion
  CTCAE
adverse events | 9 month after inclusion
  CTCAE
adverse events | 12 month after inclusion
  CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Aurore DOUGE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France